CLINICAL TRIAL: NCT03888820
Title: The Effect of Biofreeze® vs. a Placebo on Chronic Low Back Pain Walking Gait Characteristics and Pain
Brief Title: Biofreeze® vs. a Placebo on Chronic Low Back Pain Walking Gait Characteristics and Pain
Status: Active, not recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Sport and Spine Rehab Clinical Research Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: BFvP cLBP walking
Record Dates: First submitted 2018-07-09; First posted 2019-03-25 (Actual); Last update posted 2019-03-25 (Actual); Status verified 2019-03

CONDITIONS: Chronic Low Back Pain

STUDY DESIGN:
Intervention Model Description: Participants will be randomly assigned 1 of 2 topicals, Gel A or Gel B. Upon completion of study procedures they will return for a second testing session and receive the other topical
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: The participant, investigator, and statistician will be blind to the intervention received
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Biofreeze (Experimental): The Biofreeze® gel will contain 3.5% menthol while the placebo will be the same formula with menthol removed and a menthol fragrance added so it is non-distinguishable from the real Biofreeze® gel. The dose of both gels will be 5 mL applied to low back, which is consistent with previous studies who reported a treatment effect for topical gels containing menthol (1 mL of gel for every 200 cm2 of surface area). The treatment will be applied by the investigator using a gloved hand and syringe containing 5mL of gel. The gel will be applied to the low back from the lower ribs to the SI joint and iliac crests. The participant will wait 15 minutes, rate the pain in their low back.
  Interventions: Drug: Biofreeze
- Placebo (Sham Comparator): The Biofreeze® gel will contain 3.5% menthol while the placebo will be the same formula with menthol removed and a menthol fragrance added so it is non-distinguishable from the real Biofreeze® gel. The dose of both gels will be 5 mL applied to low back, which is consistent with previous studies who reported a treatment effect for topical gels containing menthol (1 mL of gel for every 200 cm2 of surface area). The treatment will be applied by the investigator using a gloved hand and syringe containing 5mL of gel. The gel will be applied to the low back from the lower ribs to the SI joint and iliac crests. The participant will wait 15 minutes, rate the pain in their low back.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Biofreeze — Biofreeze is a topical analgesic that uses the cooling effect of menthol, a natural pain reliever, to soothe minor muscle and joint pain. The product will be applied immediately after walking. The participant will wait 15 minutes prior to walking again.
  Arms: Biofreeze
Drug: Placebo — The placebo is the Biofreeze product with all active ingredients removed. The product will be applied immediately after walking. The participant will wait 15 minutes prior to walking again.
  Arms: Placebo

SUMMARY:
The purpose of this study is to determine the effect of Biofreeze® versus a placebo on walking gait characteristics and pain during walking in individuals with cLBP.

DETAILED DESCRIPTION:
A convenience sample of 20 participants, 18 years or older with cLBP will be recruited for this study. Participants must have cLBP and be able to perform all study procedures. All interested participants will report in comfortable clothing and sneakers. After explanation of the study and consent, participants will complete the demographics questionnaire, NIH cLBP Minimal Dataset, 10-point Numeric Pain Rating Scale (NPRS), and the Roland-Morris Low Back Pain and Disability Questionnaire (RMDQ). Participants will then complete a 3-minute walking baseline assessment. Following the assessment, participants will rate their pain and be randomly assigned receive a blinded topical of either Biofreeze® or a Placebo. Both the participant and the investigator will be blind to assigned products. The dose of both gels will be 5 mL per side of the low back. The participant will wait 15 minutes, rate their pain, and repeat the 3-minute walking assessment and rate their pain again. Next, there will be a minimum of a 24-72-hour washout period at which time the participants will return and repeat the same protocol using the other topical.

ELIGIBILITY:
Inclusion Criteria:

* must have cLBP and be able to perform all study procedures. CLBP will be defined as pain, muscle tension, or stiffness localized between the lower posterior margin of the rib cage and the horizontal gluteal fold lasting at least 12 weeks and has resulted in pain on at least half the days in the past 6 months

Exclusion Criteria:

* pregnancy, cancer, spinal or hip surgery, or a corticosteroid injection within the past 4 weeks

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2018-03-01 (Actual); Primary Completion 2019-03-30 (Estimated); Study Completion 2019-04-30 (Estimated)

PRIMARY OUTCOMES:
Change in Numeric Pain Rating Scale | Pain will be measured at baseline, immediately following the 3 minute walk, 15 minutes after topical application, and after the second 3 minute walk for both topical applications
  Pain will be measures on a scale of 0 to 10, 0 being no pain at all and 10 representing the worst imaginable pain.
Change in Knee Flexion | Knee Flexion Range of Motion will be measured for both topical applications at initial walk (T1) and post-topical walk (T2) in one session, lasting 30 minutes
  Knee Flexion Range of Motion will be measured using the Woodway Walker View Treadmill which utilizes a 3D camera and will be measured during the last 30 seconds of the 3 minute walk.
Change in Hip Flexion | Hip Flexion Range of Motion will be measured for both topical applications at initial walk (T1) and post-topical walk(T2), in one session, lasting 30 minutes
  Hip Flexion Range of Motion will be measured using the Woodway Walker View Treadmill which utilizes a 3D camera and will be measured during the last 30 seconds of the 3 minute walk.
Change in Step Length | Step length will be measured for both topical applications at initial walk (T1) and post-topical walk (T2), in one session, lasting 30 minutes
  Step Length will be measured using the Woodway Walker View Treadmill which utilizes load cells within the treadmill belt and will be measured during the last 30 seconds of the 3 minute walk.

CONTACTS AND LOCATIONS:
Locations (1):
- Sport and Spine Rehab, Rockville, Maryland, United States

IPD SHARING:
Plan to Share IPD: No